CLINICAL TRIAL: NCT06631690
Title: Effect of ACL Reconstruction Using Peroneus Longus Versus Hamstring Autografts on Biomechanical Properties of Ankle Joint Complex
Brief Title: Effect of ACL Reconstruction in Biomechanical Properties of Ankle Joint Complex
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Lena Mahmoud Abo Alfotoh ELbadawy, Demonstrator of Department of Biomechanics Faculty of Physical Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: P.T.REC/012/005015
Record Dates: First submitted 2024-03-18; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Anterior Cruciate Ligament Tear; Ankle Sprains
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Ankle Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Peroneus longus autograft group (Active Comparator): * Isokinetic dynamometer is a three multi-joint testing and rehabilitation device. It will be used to measure concentric peak torques of ankle planter flexor and eccentric peak torque of evertor
  * The modified Star Excursion Balance Test will be used to evaluate the dynamic balance with a series of unilateral balance tests
  * Single leg Stance (SLS) test to assess balance, especially when performed in a static position
  Interventions: Other: Isokinetic and functional balance tests
- hamstring autograft group (Active Comparator): * Isokinetic dynamometer is a three multi-joint testing and rehabilitation device. It will be used to measure concentric peak torques of ankle planter flexor and eccentric peak torque of evertor
  * The modified Star Excursion Balance Test will be used to evaluate the dynamic balance with a series of unilateral balance tests
  * Single leg Stance (SLS) test to assess balance, especially when performed in a static position
  Interventions: Other: Isokinetic and functional balance tests

INTERVENTIONS:
Other: Isokinetic and functional balance tests — Isokinetic and functional balance tests

SUMMARY:
BACKGROUND:

Anterior cruciate ligament (ACL) is an important ligamentous structure in the knee joint which contributes in maintaining stability. ACL injury contribute to approximately 50% of knee injuries .The incidence of ACL ruptures is estimated to be between 30 and 78 per 100,000 people per year .

The incidence of ACL ruptures varies depending on a number of factors, including age, sex, sport participation, and genetics. ACL ruptures are most common in young adults, particularly women. The risk of an ACL rupture has been reported as 2-8 times higher for women than for men. A systematic review study found that the risk of ACL injury was highest in football, followed by soccer, basketball, and skiing .

Nowadays, Peroneus longus tendon (PLT) autograft is used in orthopaedic surgeries. Some studies reported that PLT graft had maintained a possible more efficient ACL substitute for its tensile strength and regeneration ability after being inserted post-surgery . The PLT graft has additional benefit as it does not cause secondary injury to the knee and its adjacent structures .

Ankle proprioception is one of the crucial components contributing to postural control . PLT graft for ACL reconstruction might affect the already compromised body balance by influencing postural stability and ankle stability at the donor ankle site. So, this study will be conducted to assess and compare the effect of ACLreconstruction with PLT graft to the effect of ACL reconstruction with HT graft on ankle stability and postural control .

DETAILED DESCRIPTION:
PURPOSE

* To assess the effect of ACL reconstruction with Peroneus longus tendon autograft on Peak torque of ankle plantarflexors and evertors , Single Leg Stance test time and Star Excursion Balance Test score in patients with ACL reconstruction.
* To assess the effect of ACL reconstruction with Hamstring tendon autograft on Peak torque of ankle plantarflexors and evertors , Single Leg Stance test time and Star Excursion Balance Test score in patients with ACL reconstruction.
* To compare between the effect of ACL reconstruction with Peroneus longus tendon autograft to ACL reconstruction with Hamstring tendon autograft on peak torque of ankle plantarflexors and evertors , Single Leg Stance test time and Star Excursion Balance Test score in patients with ACL reconstruction.

HYPOTHESES

* There will be no significant effect of ACL reconstruction with Peroneus longus tendon autograft on Peak torque of ankle plantarflexors and evertors , Single Leg Stance test time and Star Excursion Balance Test score in patients with ACL reconstruction.
* There will be no significant effect of ACL reconstruction with Hamstring tendon autograft on Peak torque of ankle plantarflexors and evertors , Single Leg Stance test time and Star Excursion Balance Test score In patients with ACL reconstruction.
* There will be no significant difference in Peak torque of ankle plantarflexors and evertors , Single Leg Stance Test time and Star Excursion Balance Test score between ACL reconstruction with Peroneus longus tendon autograft and ACL reconstruction with Hamstring tendon autograft.

RESEARCH QUESTION::

* Will there be any effect of ACL reconstruction with Peroneus longus tendon autograft on Peak torque of ankle plantarflexors and evertors , Single Leg Stance test time and Star Excursion Balance Test score in patients with ACL reconstruction?
* Will there be any effect of ACL reconstruction with Hamstring tendon autograft on Peak torque of ankle plantarflexors and evertors , Single Leg Stance test time and Star Excursion Balance Test score in patients with ACL reconstruction ?
* Will there be any difference in Peak torque of ankle plantarflexors and evertors , Single Leg Stance test time and Star Excursion Balance Test score between ACL reconstruction with Peroneus longus tendon autograft and ACL reconstruction with Hamstring tendon autograft?

ELIGIBILITY:
Inclusion Criteria:

* Age ranging between 15- 45 years
* Having unilateral isolated ACL tear with no concomitant tear of other ligaments of the knee
* Having no evidence of meniscal repair
* Having bilateral healthy ankle before surgery.

Exclusion Criteria

* Pre-existing ankle injury or ankle instability
* Associated ligament injury, chondral damage, meniscal injury, fracture around the knee, and presence of pathologic condition in the lower extremity or an abnormal contralateral knee joint.
* Visible mal-alignments in the lower extremities.
* Previous surgery to the affected knee.

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-12-10 (Actual); Primary Completion 2024-04-10 (Actual); Study Completion 2024-12-10 (Estimated)

PRIMARY OUTCOMES:
Peak torque of plantarflexors and evertors (N.m) | preoperative /3 months / 6 months
  The isokinetic strength of ankle muscles will be evaluated at angular velocities of 30°/s and 120°/s in concentric/concentric mode for the ankle Planter flexion/dorsiflexion and in concentric/eccentric reciprocal action for the ankle eversion/eversion
Star Excursion Balance Test distance (cm) | preoperative /3 months / 6 months
  The Modified version of the Star Excursion Balance Test with only three directions (anterior, posterolateral [PL], and posteromedial [PM]) will be used .
  The patient will be given four practice trials to familiarize themselves with the task, followed by a brief rest. Then, three trials will be recorded with at least 10 seconds of rest between each trial. The average of the three trials will be normalized to the participant's leg length and used for analysis.
Single leg stance time (sec) | preoperative /3 months / 6 months
  The procedure will be repeated three times

CONTACTS AND LOCATIONS:
Overall Officials: Lamyaa Kotb Elsayad, PHd, Study Director — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided